CLINICAL TRIAL: NCT05119959
Title: Zambia Infant Cohort Study - Brains Optimized for Surviving and Thriving
Acronym: ZICS-BOOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-42282
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Child Development
Keywords: Children exposed to HIV in-utero but uninfected (CHEUs); Early childhood developmental (ECD) interventions; Community health workers; Home visits; Zambia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1- CHEU + ECD intervention (Experimental): Participants randomized to this arm will receive a bi-weekly community health worker-delivered ECD intervention for CHEUs
  Interventions: Other: ECD intervention for CHEUs
- Arm 2- CHEU without ECD intervention (Active Comparator): Participants randomized to this arm will receive the current Ministry of Health (MoH) standard of care with no formalized routine assessment of neurodevelopment.
  Interventions: Other: Usual care for CHEUs
- Arm 3- HIV Unexposed (HUU) without ECD intervention (Active Comparator): Participants randomized to this arm will receive the current Ministry of Health (MoH) standard of care with no formalized routine assessment of neurodevelopment.
  Interventions: Other: Usual care for CHEUs

INTERVENTIONS:
Other: ECD intervention for CHEUs — The bi-weekly community health worker-delivered ECD 1 hour intervention using the modules from the SUPERCDZ curriculum which is a Zambian adaptation of UNICEF's Nurturing Care Framework
  Arms: Arm 1- CHEU + ECD intervention
Other: Usual care for CHEUs — No ECD interventions will be provided by community health workers. Children will be followed at clinics for growth and monitoring, vaccinations on a MoH approved schedule.
  Arms: Arm 2- CHEU without ECD intervention; Arm 3- HIV Unexposed (HUU) without ECD intervention

SUMMARY:
Children exposed to HIV in-utero but uninfected (CHEUs) number 14.8 million globally. In Zambia, an estimated 56,000 CHEUs are born annually, a staggering fraction of the national birth cohort. Multiple studies establish that CHEUs are more neurodevelopmentally vulnerable than HIV-unexposed peers. In Zambia, there are existing effective early childhood developmental (ECD) interventions that target other vulnerable populations, but never trialed specifically for CHEUs. Scaling up ECD is now a priority of Zambia's national strategy, but CHEUs are not currently targeted.

There is a need to better understand the scope and mechanism of CHEU-related neurodevelopmental differences and what interventions are most effective. This randomized clinical trial (RCT) is a true effectiveness trial as the intervention will deploy a home-based adaptation of the same curriculum that is currently used elsewhere in the country, named Scaling Up Early Childhood Development In Zambia (SUPERCDZ). The effectiveness of a scalable early childhood development (ECD) intervention for CHEUs will be evaluated using normalized Z-scores of neurodevelopmental testing at age 24 months.

In this RCT the investigators will test the following hypotheses:

Hypothesis 1: An ECD intervention delivered by community health workers via bi-weekly home visits will improve neurodevelopmental outcomes in CHEUs.

Hypothesis 2: CHEUs have significantly worse neurodevelopmental outcomes than unexposed peers at 24 months, mediated by preterm birth, disease stage or antiretroviral (ARV) exposure.

This RCT will build on an existent, actively recruiting cohort of 1500 pregnant women-infant dyads in a peri-urban hospital in Zambia, the Zambian Infant Cohort Study (ZICS), by extending the follow-up of a subsample of infants from 6 months to 2 years amongst the last 525 children enrolled (ZICS-BOOST- Brains Optimized to Survive and Thrive). The study will have three arms: Arm 1) CHEU + ECD intervention (n=175); Arm 2) CHEU without ECD intervention (n=175); Arm 3) HUU without intervention (n=175).

ELIGIBILITY:
Inclusion Criteria:

* Zambia Infant Cohort Study (ZICS) cohort participants who are >18 years old AND are still pregnant OR whose infants are less than 9 months of age by February 2022.
* ZICS inclusion criteria were pregnant women (1:1, HIV+:HIV-) presenting for antenatal care at Chawama First Level Hospital and intending to deliver at Chawama First Level Hospital and less than 26 weeks gestation by ultrasound

Exclusion Criteria:

* Mother-infant dyads not enrolled in ZICS
* Mother-infant dyads where mother is <18 years of age

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 469 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Neurodevelopment at 18 months post enrollment | 18 months
  The Malawi Developmental Assessment Tool (MDAT) will be used to assess neurodevelopment. MDAT provides an independent evaluation of development in the domains of gross motor, fine motor, language and social skills. The MDAT can be administered in any environment as it requires minimal equipment and is more culturally relevant to our context. The scores from the MDAT are relatable and comparable to those obtained from the Bayley Scales of Infant and Toddler Development 3rd Edition (BSID-III). Primary outcomes will be z-scores from four neurodevelopmental domain measurements-gross motor, fine motor, language, and social.

SECONDARY OUTCOMES:
Neurodevelopment at 6 months post enrollment | 6 months
  The Malawi Developmental Assessment Tool (MDAT) will be used to assess neurodevelopment. MDAT provides an independent evaluation of development in the domains of gross motor, fine motor, language and social skills. The MDAT can be administered in any environment as it requires minimal equipment and is more culturally relevant to our context. The scores from the MDAT are relatable and comparable to those obtained from the BSID-III. Primary outcomes will be z-scores from four neurodevelopmental domain measurements-gross motor, fine motor, language, and social.
Language development at 6, 12, and 18 months post enrollment | 6 months. 12 months, 18 months
  Children's language development will be assessed at 12 and 24 months using an adapted MacArthur-Bates Communicative Development Inventories (CDI) tool.
Child's age-specific tasks at 6, 12, and 18 months post enrollment | 6 months, 12 months, 18 months
  The Caregiver Reported Early Development Instrument (CREDI) will be used to assess age-specific tasks for early childhood 0-36 months. It is intended to be used at a population level to detect developmental delay, not as an individual diagnostic tool. This open-source, psychometrically sound tool has been tested in over 15 low-and-middle-income countries and is culturally and linguistically neutral. When deployed in its long form it can be analyzed by specific developmental domains including (motor, language and cognitive, socio-emotional). CREDI scores per arm will be described in z-scores from four neurodevelopmental domain measurements.
Caregiver mental health and wellbeing at 6, 12 and 18months post enrollment | 6 months, 12 months, 18 months
  The Self-Reporting Questionnaire 20 (SQR-20) will be used to assess Caregiver mental health and wellbeing. The SQR-20 has 20 questions that assess for common mental health conditions and common physical manifestations of depression or anxiety (e.g., poor appetite, poor sleep, anhedonia). There are 20 questions and more yes answers correlate with higher risk for mental health concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Herlihy, MD MPH, Principal Investigator — BU School of Public Health; Ethan Zulu, MBChB MSc, Principal Investigator — Right to Care - Zambia
Locations (2):
- Boston University School of Public Health, Boston, Massachusetts, United States
- Right to Care Zambia, Lusaka, Longacres, Zambia

IPD SHARING:
Plan to Share IPD: No